CLINICAL TRIAL: NCT01305850
Title: The Effect of Aliskiren and Losartan on Peritoneal Membrane in Continuous Ambulatory Peritoneal Dialysis Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Assist. Prf. Talerngsak Kanjanabuch, M.D / Department of nephrology, Division of Internal medicine, Faculty of medicine, Chulalongkorn University, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 162/53
Record Dates: First submitted 2010-11-30; First posted 2011-03-01 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-02

CONDITIONS: Peritoneal Membrane Failure
Keywords: Aliskiren; Losartan; Peritoneal membrane dysfunction
MeSH Terms: interventions — aliskiren; Losartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Aliskiren (Active Comparator)
  Interventions: Drug: Aliskiren
- Aliskiren plus Losartan (Active Comparator)
  Interventions: Drug: Aliskiren plus Losartan
- Enalapril plus Losartan (Active Comparator)
  Interventions: Drug: Enalapril plus Losartan
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Patients in the control group will administer antihypertensive agents, except angiotensin converting enzyme inhibitors, angiotensin receptor blockers and spironolactone. Dosages are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Control
  Arms: placebo
Drug: Aliskiren — Patients with hypertension will take fixed-dose 150 mg aliskiren per day. Antihypertensive agents other than angiotensin converting enzyme inhibitors, angiotensin receptor blocker and spironolactone will be allowed and dosages are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Aliskiren group
  Arms: Aliskiren
Drug: Aliskiren plus Losartan — Patients with hypertension will take fixed-dose 150 mg aliskiren + 50 mg losartan per day. Antihypertensive agents other than angiotensin converting enzyme inhibitors, angiotensin receptor blockers and spironolactone will be allowed and dosages are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Aliskiren plus Losartan group
  Arms: Aliskiren plus Losartan
Drug: Enalapril plus Losartan — Patients with hypertension will take fixed-dose 20 mg enalapril + 50 mg losartan per day. Antihypertensive agents other than angiotensin converting enzyme inhibitors, angiotensin receptor blockers and spironolactone will be allowed and dosages are adjusted appropriately to achieve and maintain the target blood pressure of 130/80 mmHg
  Other Names: Enalapril plus Losartan group
  Arms: Enalapril plus Losartan

SUMMARY:
This is a prospective, randomized, placebo controlled, multi-center clinical trial to determine whether aliskiren or aliskiren plus losartan or enalapril plus losartan effects on peritoneal membrane transportation.

DETAILED DESCRIPTION:
Detailed description:

Many peritoneal dialysis patients suffer from uremia due to inadequate dialysis or volume overload caused by failure of peritoneal membrane transportation. One of the most important etiologies of peritoneal membrane failure is unavoidable to use high glucose-containing dialysate solution that induces injury to mesothelial cells. Previous data found that injured mesothelial cell produced Angiotensin II inducing peritoneal inflammation and fibrosis. Blockade of the renin-angiotensin system by angiotensin-converting enzyme inhibition or angiotensin receptor antagonism play a major role to slow these effects.

Many trials in animal studies have proved the benefit of angiotensin-converting enzyme inhibition and angiotensin receptor antagonism in preservation of peritoneal membrane but clinical evidences in human are controversy in the past. Recently our data have demonstrated the roles of angiotensin-converting enzyme inhibition and angiotensin receptor antagonism for slowing peritoneal membrane dysfunction in views of anatomy and solute transportation (abstract presentation in American Society of Nephrology 2010). These available data confirmed that renin-angiotensin system blockages were benefit. Nowadays, there is a new class of antihypertensive drug, called direct renin inhibitor . It blocks (pro)renin active site that is the rate- limiting step of renin-angiotensin system. We're interesting in this drug and wonder it can slow the peritoneal membrane dysfunction in continuous ambulatory peritoneal dialysis patients. Therefore, we design a study to show the effect of aliskiren alone or combination with angiotensin receptor antagonism for slowing peritoneal membrane dysfunction in naive continuous ambulatory peritoneal dialysis patients in several hospitals. Our study will be taken in 1 year duration and uses modified peritoneal equilibrium test and dialysate cancer antigen 125 (CA125) as indexes of peritoneal membrane transportations.

ELIGIBILITY:
Inclusion Criteria:

1. All patients received continuous ambulatory peritoneal dialysis less than one and a half years
2. Subjects of either sex, more than 20 years old
3. Hypertension
4. Provision of written informed consent by subject or guardian

Exclusion Criteria:

1. No history of taking an angiotensin converting enzyme inhibitor or angiotensin-receptor blockers or aldosterone antagonist for at least 2 month
2. Serum potassium more than 5.5 mEq/L
3. History of renal artery stenosis
4. Peritonitis or volume overload within the preceding 1 month
5. Myocardial infarction within the preceding 6 months or clinically significant valvular disease or any active cardiovascular disease
6. History of malignant hypertension or hypertensive encephalopathy or cerebrovascular accident within the preceding 6 months
7. Any condition that may have precluded a patient from remaining in the study, such as alcohol or drug abuse, chronic liver disease, malignant disease, or psychiatric disorder
8. History of allergy or intolerance to an angiotensin converting enzyme inhibitors or angiotensin receptor blockers
9. Hypotension defined as systolic blood pressure less than 90 mmHg

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Changing in modified peritoneal equilibrium test | at the beginning, 6 months and 12 months
  Modified peritoneal equilibrium test is the standard test for evaluation peritoneal membrane transportation.

SECONDARY OUTCOMES:
appearance rate of dialysate CA125 | the begining, 6 months and 12 months
  Appearance rate of dialysate CA125 refers to anatomical change of peritoneal. It can be calculated by multiplying dialysate CA125 with dialysate volume and deviding by dwell time.
nutritional status | at the beginning, 6 months and 12 months
  assess by serum albumin and subjective global assessment
adverse events | 12 months
  adverse events of the drugs

CONTACTS AND LOCATIONS:
Overall Officials: Talerngsak Kanjanabuch, Assist. Prf., Principal Investigator — Investigator; Pichaya Tantiyavarong, MD., Study Director — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand